CLINICAL TRIAL: NCT04364347
Title: Chemotherapy-induced Circadian Rhythm Disruption: Investigation Using Biomarker
Brief Title: Chemotherapy-induced Circadian Rhythm Disruption
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Other Study IDs: CIRCADIAN
Record Dates: First submitted 2020-04-21; First posted 2020-04-28 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Breast Neoplasms
Keywords: Breast neoplasms; Circadian rhythm; Chemotherapy; Biomarker; Core body temperature; Melatonin; Cortisol; Circadian gene
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate chemotherapy-induced circadian rhythm disruption through biomarkers, and the relationship between chemotherapy-induced circadian rhythm disruptions and side effects of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Those who have undergone breast cancer surgery and are waiting for chemotherapy
2. premenopausal women
3. Invasive adenocarcinoma of the breast stages I-III

Exclusion Criteria:

1. Other cancer diagnosis within the last 5 years
2. Other physical problems that can affect survival
3. Other physical problems that can affect sleep or mood ex) pulmonary disease(COPD, Asthma), GI disorder(GERD), Renal disorder(End stage renal disease), Endocrine disorder(Hypothyroidism, Acromegaly), Infectious disease(Viral, bacterial infections, HIV infections), Neurological disease(epilepsy, parkinson's disease, neuromuscular disorder, stroke, multiple sclerosis), Cardiovascular disease(Coronary heart disease), Pain, etc.
4. ECOG(Eastern Cooperative Oncology Group performance status) >1
5. In the case of depression, anxiety disorder, sleep disorder, etc.
6. If you have worked night shifts or shifts within the past 6 months
7. Weight 40kg or less, digestive diseases, history of gastrointestinal surgery, etc.
8. If you are currently taking psychiatric drugs (antipsychotics, antidepressant, mood stabilizer, benzodiazepine, psychostimulant, beta-blocker, etc.)
9. If you have traveled on a transmeridian plane in the 3rd zone or more within the past 6 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: University (Tertiary) hospital, oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2019-12-14 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma melatonin, cortisol levels before, after and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), T2(9 months after chemotherapy termination)
  12 times in 24 hours at 2 hour intervals
Changes in core body temperature before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), T2(9 months after chemotherapy termination)
  for 24 hours
Changes in PBMC(Peripheral Blood Mononuclear Cell) mRNA levels before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), T2(9 months after chemotherapy termination)
  12 times in 24 hours at 2 hour intervals
Changes in plasma protein levels before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  6 times in 24 hours at 4 hour intervals
DNA | T0(2 weeks before the start of chemotherapy)
  First one only

SECONDARY OUTCOMES:
Changes in MAT scores before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  MAT(Multinational Association of Supportive Care in Cancer Antiemesis tool) / Evaluating acute/delayed nausea and vomiting in patients treated with chemotherapy / High scores mean severe nausea and vomiting
Changes in EORTC-QLQ CIPN20 scores before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  EORTC-QLQ CIPN20(European Organization for Research and Treatment of Cancer Quality of Life Chemotherapy-induced Peripheral Neuropathy) / Peripheral neuropathy evaluation (It consists of 9 questions of sensory nerve area, 8 questions of motor nerve area and 3 questions of autonomic nerve area.) / High scores mean severe peripheral neuropathy
Changes in Hot flush symptoms before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  Assessment of the number and severity of hot flashes (mild, moderate, severe) for 1 week / High scores mean severe hot flush
Changes in MEQ scores before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  MEQ(Morningness-Eveningness Questionnaire) / Individual circadian rhythm evaluation / Consists of 19 questions
Changes in MCTQ scores before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  MCTQ(Munich Chronotype Questionnaire) / Assessment of circadian rhythm discrepancies
Changes in FACT-B scores before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  FACT-B(Functional Assessment of Cancer Therapy-Breast) / Measuring the quality of life of breast cancer patients / Self-report questionnaire of 44 items / High score means low quality of life
Changes in MDASI scores before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  MDASI(M. D. Anderson Symptom Inventory) / Cancer-related physical symptoms evaluation / High score means severe physical symptoms
Changes in HADS scores before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  HADS(Hospital anxiety and depression scale) / Depression, anxiety evaluation of patients with physical illness / Self-report questionnaire with 14 items / High score means severe depression and anxiety symptoms
Changes in MSPSS scores before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  MSPSS(Multidimensional Scale of Perceived Social Support) / Social support assessment / Self-report questionnaire of 12 items / High score means high social support
Changes in PSQI scores before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  PSQI(Pittsburgh Sleep Quality Index) / Evaluate sleep quality in the past month / High scores mean severe sleep disorders
Changes in Actigraphy pattern before chemotherapy, after chemotherapy, and 9 months after chemotherapy | T0(2 weeks before the start of chemotherapy), T1(2 weeks after chemotherapy termination), C3(Just before the third chemotherapy), C7(Just before the 7th chemotherapy), T2(9 months after chemotherapy termination)
  Activity measurement / Records information such as weekly activity, time to go to bed, sleep incubation period, number of awakenings during sleep, wake-up time, and brightness of ambient light

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Jin Hahm, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

REFERENCES:
- [Derived] Shin JS, Jung S, Won GH, Lee SH, Kim J, Jung S, Yeom CW, Lee KM, Son KL, Kim JI, Jeon SY, Lee HB, Hahm BJ. The Association Between Circadian Disruption in Core Body Temperature Rhythm and Post-Chemotherapy Sleep Disturbances in Breast Cancer Survivors. J Sleep Res. 2025 Apr 29:e70080. doi: 10.1111/jsr.70080. Online ahead of print. PMID 40296750
- See also: study site webpage — http://www.snuh.org/
- See also: Institutional Review Board — https://cris.snuh.org/ncris/